CLINICAL TRIAL: NCT05646225
Title: Effects of Early Mobilization With and Without Chest Physiotherapy on Dyspnea, Pulmonary Function Test and Quality of Life in Elderly Patients With Chronic Bronchitis.
Brief Title: Early Mobilization With and Without Chest Physiotherapy in Chronic Bronchitis Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0315 Mishal Tanveer
Record Dates: First submitted 2022-11-24; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Chronic Bronchitis
Keywords: early mobilization, chest physiotherap, chronic bronchitis
MeSH Terms: conditions — Bronchitis, Chronic | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chest physiotherapy and early mobilization (Experimental): Chest Physiotherapy: Each session included a series of exercises, lasting a total of 15 minutes and including positioning,self-conscious breathing control, diaphragmatic breathing control, and exercises for the chest wall and abdominal muscle walls.
  Early mobilization: Each session included abdominal and upper and lower limb exercises, shoulder and full arm circling, lying to sit, sit to stand, walk and other exercises. This training has been described previously and used in other clinical trials. Each exercise was repeated 8-10 times over 30 minutes
  Interventions: Other: chest physiotherapy and early mobilization; Other: early mobilization
- early mobilization (Active Comparator): Each session included abdominal and upper and lower limb exercises, shoulder and full arm circling, lying to sit, sit to stand, walk and other exercises. This training has been described previously and used in other clinical trials. Each exercise was repeated 8-10 times over 30 minutes.
  Interventions: Other: early mobilization

INTERVENTIONS:
Other: chest physiotherapy and early mobilization — Chest Physiotherapy: Each session included a series of exercises, lasting a total of 15 minutes and including positioning self-conscious breathing control, diaphragmatic breathing control, and exercises for the chest wall and abdominal muscle walls.
  Early mobilization: Each session included abdominal and upper and lower limb exercises, shoulder and full arm circling, lying to sit, sit to stand, walk and other exercises. This training has been described previously and used in other clinical trials. Each exercise was repeated 8-10 times over 30 minutes
  Arms: chest physiotherapy and early mobilization
Other: early mobilization — Each session included abdominal and upper and lower limb exercises, shoulder and full arm circling, lying to sit, sit to stand, walk and other exercises. This training has been described previously and used in other clinical trials. Each exercise was repeated 8-10 times over 30 minutes

SUMMARY:
It will be a randomized control trial study in which data are collected from hospital. A sample of 26 patients will divided into two group. One group of 13 patients will receive early mobilization and other group of 13 patients will receive early mobilization and chest physiotherapy only. All subject will receive 30 minute two session per day till two weeks. Outcome will be measured with MRC dyspnea scale and Pulmonary function test with spirometry to measure FEV1 and FEV1/FVC and quality of life will be checked by using ST. GEORGE'S respiratory questionnaire. Data will be analyzed by using SPSS version 21.

DETAILED DESCRIPTION:
It will be a randomized control trial study in which data are collected from Jinnah hospital Lahore. A sample of 26 patients will be included and divided into two group. One group of 13 patients will receive early mobilization with chest physiotherapy and other group of 13 patients will receive early mobilization only. All subject will receive 30 minute two session per day till two weeks. Outcome will be measured with MRC dyspnea scale and Pulmonary function test with spirometry to measure FEV1 and FEV1/FVC and quality of life will be checked by using ST. GEORGE'S respiratory questionnaire. Data will be analyzed by using SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Both gender of age 45-70 years
* Patient diagnosed with chronic bronchitis (admitted patients)
* Taking bronchodilators

Exclusion Criteria:

* • Patient having any other condition cardiovascular, diabetes mellitus and neurological conditions

  * Patient history of radiotherapy
  * Unconscious ICU patients
  * Patient received any pre-admitted Physiotherapy protocol

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
St. George Respiratory Questionnaire | Two weeks
  Using the SGRQ-C, the QOL of the study participants is evaluated. There are 14 questions in this questionnaire. The questionnaire would be given to the patients, who will instructed to answer it truthfully. The response is whatever they believe to be true for them. The minimum and maximum values are 0 and 100, respectively. Better QOL is indicated by a lower score. The formula was used to determine the total of the three component scores (symptoms, activity, and effects).

OTHER OUTCOMES:
pulmonary function test FEV1 | Two weeks
  spirometery is portable, and handheld device used to measure capacities and volumes of lungs. predicted percentage(%) value of FEV1. The patient stands up straight, then takes a deep breath, and holds it till the mouthpiece is placed in between the teeth. Instruct the patient not to put the tongue against or inside the hole of the mouthpiece. The patient was asked to blow in the hole as fast and hard in a single blow. The first burst of air is the most important. The number was noted down, and the same procedure was repeated three times. The best of the three readings was the value used for the analysis. evaluation will be done before and after 2 week treatment plan
pulmonary function test | Two weeks
  spirometery is portable, and handheld device used to measure capacities and volumes of lungs. predicted percentage(%) value of FEV1/FVC will be recorded through spirometery. The patient stands up straight, then takes a deep breath, and holds it till the mouthpiece is placed in between the teeth. Instruct the patient not to put the tongue against or inside the hole of the mouthpiece. The patient was asked to blow in the hole as fast and hard in a single blow. The first burst of air is the most important. The number was noted down, and the same procedure was repeated three times. The best of the three readings was the value used for the analysis. evaluation will be done before and after 2 week treatment plan
MRC dyspnea scale | Two weeks
  Using the MRC dyspnea scale, self-perceived dyspnea in connection to physical impairment has been evaluated. Patients is required to rate their self-perceived dyspnea on a scale of (0-4) using pre-defined sentences. There will be pre- and post-treatment evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha younas, MS, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No